CLINICAL TRIAL: NCT01386567
Title: A One Year Open Label Study of Androxal in the Treatment of Secondary Hypogonadism in Men Who Have Completed Protocol ZA-203
Brief Title: A One Year Open Label Study for the Treatment of Hypogonadism (Low Testosterone) in Men Who Have Completed ZA-203
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Repros Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZA-203 Extension
Record Dates: First submitted 2011-06-29; First posted 2011-07-01 (Estimated); Last update posted 2013-05-17 (Estimated); Status verified 2013-05

CONDITIONS: Hypogonadism; Low Testosterone
Keywords: hypogonadism; low testosterone; low T
MeSH Terms: conditions — Hypogonadism | interventions — Enclomiphene; Testosterone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Androxal (Experimental): Androxal (enclomiphene citrate)12.5 mg or 25 mg
  Interventions: Drug: Androxal (enclomiphene citrate)
- Testim (topical testosterone) (Active Comparator)
  Interventions: Drug: Testim (topical testosterone)

INTERVENTIONS:
Drug: Androxal (enclomiphene citrate) — capsules oral 1x a day
  1 year
  Other Names: enclomiphene citrate
  Arms: Androxal
Drug: Testim (topical testosterone) — topical
  1 tube
  1x a day
  1 year
  Other Names: topical testosterone; exogenous testosterone; testosterone gel
  Arms: Testim (topical testosterone)

SUMMARY:
The purpose of this study is to determine the continued effects of Androxal on morning testosterone and reproductive status in men with secondary hypogonadism who have completed protocol ZA-203. Men will be allowed to choose Androxal (enclomiphene citrate) or Testim (topical testosterone) at the beginning of the study. All men on Androxal will start at 12.5 mg and will be allowed to up titrate to 25 mg if an inadequate response is exhibited at the lower dose.

ELIGIBILITY:
Inclusion Criteria:

* Successful completion of ZA-203
* Ability to understand and provide written informed consent
* Agreement to use a condom, and with a fertile female partner, another form of contraception
* Agreement to provide semen samples in the clinic

Exclusion Criteria:

* Any condition which, in the opinion of the Investigator, would make the Subject an unsuitable candidate for enrollment in the study

Ages: 21 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2011-07; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Change in testosterone comparing Androxal to Testim | 1 year
  Values of total morning testosterone levels at each visit comparing Androxal (enclomiphene citrate) 12.5 and 25 mg and Testim

SECONDARY OUTCOMES:
Change in leuteinizing hormone and follicle stimulating hormone comparing Androxal (enclomiphene citrate) to Testim (topical testosterone) | 1 year
  Values of follicle stimulating hormone (FSH) and leuteinizing hormone (LH) at each visit comparing Androxal 12.5 and 25 mg to Testim
Changes in sperm parameters from baseline comparing Androxal (enclomiphene citrate) to Testim (topical testosterone) | 1 year
  Reproductive safety will be assessed by changes in values from baseline of semen volume, and sperm concentration, total count, morphology and motility at baseline (Visit 1), month 4, 6 and 12 comparing Androxal 12.5 and 25 mg to Testim

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Garden Grove, California
  - Sacramento, California
  - San Diego, California
  - Las Vegas, Nevada
  - Houston, Texas

REFERENCES:
- See also: Sponsor website — http://www.reprosrx.com
- See also: Study information — http://helpmylowT.com